CLINICAL TRIAL: NCT02372695
Title: Effect of Paricalcitol Over Vessel Wall: Pleiotropic Analogues Vitamin D Effects
Brief Title: Effect of Paricalcitol Over Vessel Wall
Acronym: MICROBUB
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol showed to be inappropriate for the evaluation of the selected patients
Sponsor: Effice Servicios Para la Investigacion S.L. (Industry)
Collaborators: Jaume Arnó Renal Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MICROBUB-2011-01; 2011-002554-30 (EudraCT Number)
Record Dates: First submitted 2013-03-05; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Nephropathy
MeSH Terms: conditions — Kidney Diseases | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Patient will take one pill of paricalcitol a day.
  Interventions: Drug: Paricalcitol
- Usual treatment. (No Intervention): Patient allocated to this arm will only take his/her habitual treatment

INTERVENTIONS:
Drug: Paricalcitol
  Other Names: Zemplar- 1 ug/day
  Arms: Treatment

SUMMARY:
To provide evidence based prospectives of the potential benefit effects of paricalcitol, an analog of vitamin D, over the prevention / retardation of the progression of neoangiogenesis (vessels), atherosclerosis and vascular calcification.

DETAILED DESCRIPTION:
Providing prospective results based on evidence of potential beneficial effects of paricalcitol, an analogue of vitamin D in the prevention / delay of progression of neoangiogenesis (vessels), atherosclerosis and vascular calcification.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 50 and 75 years.
* Chronic kidney disease stage 5 D or 4-5 No D as calculated glomerular filtration rate (MDRD).
* Concentration of intact parathyroid hormone (iPTH): 150-400 pg/ml.
* Plasma concentrations of 25 (OH) vitamin D <30 ng/ml.
* Without vitamin D supplementation for 3 months before the study.
* Serum P> 3.8 mg / dl.
* Serum Ca> 9.8 mg / dl.
* No history of cardiovascular events (angina or myocardial infarction, stroke, peripheral arterial disease).
* No exclusion criteria for the use of contrast.

Exclusion Criteria:

* Allergic reaction to sulfur hexafluoride.
* Recent unstable cardiac symptoms.
* Patients with recent coronary intervention (<7 days)
* Patients with class III and IV heart failure or severe arrhythmias.
* Severe pulmonary hypertension.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Prevention on vessels progression based on paricalcitol intake. | participants will be followed for the duration of whole study, an expected average of 1 year
  Providing prospective results based on evidence of potential beneficial effects of paricalcitol, an analogue of vitamin D in the prevention / delay of progression of neoangiogenesis (vessels), atherosclerosis and vascular calcification.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Vittoria Arcidiacono, Ph D, Principal Investigator — Hospital Universitario Arnau de Vilanova de Lleida.